CLINICAL TRIAL: NCT01737385
Title: Intraoperative Examination of Microcirculation of the Caput Humeri After Traumatic Proximal Humerus Fracturation.
Brief Title: Examination of Microcirculation of the Caput Humeri After Proximal Humerus Fracture
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: CTC-A10-31
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Proximal Humeral Fractures
Keywords: microcirculation; proximal humeral fractures; O2C
MeSH Terms: conditions — Shoulder Fractures | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Type 1: One segment fracture
  Interventions: Procedure: Measurement with O2C
- Type 2: Two segment fracture
  Interventions: Procedure: Measurement with O2C
- Type 3: Three segment fracture
  Interventions: Procedure: Measurement with O2C
- Type 4: Four segment fracture
  Interventions: Procedure: Measurement with O2C

INTERVENTIONS:
Procedure: Measurement with O2C — Measurement of microcirculation using O2C light probes.

SUMMARY:
This study examines the microcirculation of the caput humeri after proximal humeral fracturation using O2C light probes.

During the operation the blood circulation is measured at four points (tuberculum majus, tuberculum minus, neck and head of the humerus) directly on the bone. The O2C light probes are a none-invasive technique of measuring blood flow, velocity and oxygen concentration. The data is analysed in respect to the fracture type according to the classification of Neer.

Valuable additional information for the correct treatment and prognosis of humeral fractures is expected.

ELIGIBILITY:
Inclusion Criteria:

* traumatic fractures of the proximal humerus
* surgical treatment
* over eighteen years of age

Exclusion Criteria:

* pathological fractures
* conservative treatment
* soft tissue damage
* delay of surgery more than three days
* immunological defects
* multiple trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that are treated for proximal humeral fratures in the University hospital of the RWTH Aachen University.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
microcirculation of the caput humeri | during surgery
  oxygen saturation, haemoglobin, blood flow, velocity of blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christoph Pape, Univ.-Prof MD, Study Chair — Dpt. of Orthopedic Trauma, RWTH Aachen University
Locations (1):
- RWTH Aachen University Hospital, Aachen, Nordrheinwestfalen, Germany